CLINICAL TRIAL: NCT03632915
Title: Pharmacokinetics of Antiepileptic Drugs in Critically Ill Patients Undergoing Continuous Renal Replacement Therapy
Brief Title: Pharmacokinetics of Antiepileptics in Patients on CRRT
Acronym: PADRE
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Neeraj Badjatia, Professor of Neurology, University of Maryland, Baltimore
Other Study IDs: HP-00066222
Record Dates: First submitted 2018-07-25; First posted 2018-08-16 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Acute Kidney Injury; Renal Insufficiency; Renal Failure; Pharmacokinetics
Keywords: Antiepileptics; Continuous Renal Replacement Therapy
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency | interventions — Levetiracetam; Lacosamide; Phenytoin; Phenobarbital; Ketamine; Valproic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- No study intervention: No study intervention
  Interventions: Drug: Levetiracetam; Drug: Lacosamide; Drug: Phenytoin; Drug: Phenobarbital; Drug: Ketamine; Drug: Valproic Acid

INTERVENTIONS:
Drug: Levetiracetam — Standard of care
Drug: Lacosamide — Standard of care
Drug: Phenytoin — Standard of care
Drug: Phenobarbital — Standard of care
Drug: Ketamine — Standard of care
Drug: Valproic Acid — Standard of care

SUMMARY:
The purpose of the study is to measure levels of any of the following AEDs (levetiracetam, phenobarbital, phenytoin, ketamine, valproic acid, lacosamide) in blood and effluent on critically ill patients receiving CRRT in order to characterize drug pharmacokinetics and optimize dosing strategies in patients on CRRT.

ELIGIBILITY:
Inclusion Criteria:

* Expected to be on CRRT and receive any of the following for more than 24 hrs
* Expected to survive for more than 24 hrs
* Achievement of steady state drug concentrations prior to study enrollment

Exclusion Criteria:

* Pregnancy
* Age < 18
* Prisoner

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing CRRT who are also being treated with an antiepileptic drug
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Influence of renal replacement therapy on drug exposure (AUC of plasma concentration levels) | Single Dosing Interval - 12 hours
  Simultaneous samples will be taken from pre-filter, post-filter, and effluent sampling ports before dose administration, after the completion of the infusion or 1 hours post oral dose, and 6 additional time points post-infusion or post oral administration.
Influence of renal replacement therapy on drug clearance | Single Dosing Interval - 12 hours
  Simultaneous samples will be taken from pre-filter, post-filter, and effluent sampling ports before dose administration, after the completion of the infusion or 1 hours post oral dose, and 6 additional time points post-infusion or post oral administration.
Determination of drug specific sieving coefficient (SC) | Single Dosing Interval - 12 hours
  SC is a measure of a filter efficiency in clearing drugs and solute. SC will be calculated using pre-filter and effluent concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Badjatia, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No